CLINICAL TRIAL: NCT03418116
Title: Argus II Retinal Prosthesis System - Better Vision RP Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company Decision
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-08-01
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Argus II (Experimental): Implantation of the Argus II Retinal Prosthesis in patients with advanced Retinitis Pigmentosa who have a measurable central residual visual field smaller than or equal to 5 degrees radius. The array will be placed parafoveally, adjacent to the preserved central visual field (i.e., "tunnel vision") in these subjects.
  Interventions: Device: Argus II Retinal Prosthesis

INTERVENTIONS:
Device: Argus II Retinal Prosthesis — The Argus II System is designed to provide visual function to individuals with severe to profound vision loss due to outer retinal degeneration. It consists of implanted and external components. The implant is an epiretinal prosthesis that is surgically implanted in and around the eye. The external equipment includes glasses and a video processing unit (VPU). The glasses include a miniature video camera, which captures video images, and a coil that sends data and stimulation commands to the implant. The VPU converts the video images into stimulation commands and is body-worn. The Argus II System operates by converting video images into electrical energy that activates retinal cells, delivering the signal through the optic nerve to the brain where it is perceived as light.

SUMMARY:
The study is conducted to evaluate the safety and benefit of the Argus II System in a selected patient population with advanced Retinitis Pigmentosa who have a measurable central residual visual field smaller than or equal to 5 degrees radius.

DETAILED DESCRIPTION:
The Argus II System is intended for use in blind patients with severe to profound retinitis pigmentosa with at least some light perception in the eye to be implanted.

The majority of RP patients still have some central vision even at a very late stage of the disease. This extremely restricted visual field is, however, highly disabling in daily life. The primary objective of this study is to evaluate the safety and benefit of the Argus II System in RP patients characterized as late stage with a central residual visual field smaller than or equal to 5 degrees radius . The electrode array will be placed in a para- to peri foveal location adjacent to the subject's residual visual field, thus increasing the total retinal area receptive to light.

Safety data will be monitored to ensure continued acceptability of risks to study subjects and visual function will be measured to evaluate the effectiveness of the system in this "better vision" RP population. In addition, effects on functional vision and quality of life will be assessed through the Functional Low-Vision Observer Rated Assessment (FLORA) and the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25).

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 25 years or older;
* Diagnosed with advanced Retinitis Pigmentosa (including syndromic RP), Choroideremia, Leber's Congenital Amaurosis, or Rod-Cone disease;
* A measurable central residual visual field of 5° radius or smaller in both eyes, as determined by Goldmann perimetry;
* Visual acuity of 0.1 (1.0 logMAR) or worse in the eye to be implanted, as measured by ETDRS chart;
* Previous history of useful form vision;
* Provided written, informed consent to participate in the study.

Exclusion Criteria:

* Ocular diseases or conditions that could prevent the Argus II implant from working (e.g., optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, etc.);
* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva; axial length <20.5 mm or > 26 mm; corneal ulcers; choroidal neovascularization in the area of the intended tack location, etc.);
* Pre-disposition to eye rubbing;
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  1. cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
  2. psychiatric disease including diagnosed forms of depression;
  3. does not speak a principal language associated with the region, and
  4. deafness or selective frequency hearing loss that prevents hearing device alarms and alerts;
* Pregnant or wish to become pregnant during the course of the study;
* Participating in another investigational drug or device study that may conflict with the objectives, follow-up, or testing of this study;
* Inability to tolerate general anaesthesia or the recommended antibiotic and steroid regimen associated with the implantation surgery;
* Conditions likely to limit life to less than 1 year from the time of inclusion.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 Years
  The nature and number of adverse events in implanted subjects.
Visual field | 2 Years
  The effect of the Argus II System on visual field size, as measured by Goldmann perimetry

SECONDARY OUTCOMES:
Visual function | 2 Years
  Effect of the Argus II System on visual function, as measured by a suite of visual tests
Quality of Life | 2 Years
  Effect of the Argus II System on quality of life, as measured by the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25)
Functional vision and quality of life | 2 Years
  The general impact of the Argus II on subject's lives, as measured by the Functional Low-Vision Observer Rated Assessment (FLORA)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Walter, Prof Dr med, Principal Investigator — RWTH Aachen University
Locations (3):
- Germany (3):
  - Augenklinik Städtisches Klinikum Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - University Medical Center Schleswig-Holstein, Department of Ophthalmology, Lübeck, Schleswig-Holstein
  - RWTH University Eye Clinic, Aachen